CLINICAL TRIAL: NCT00227656
Title: Phase II Trial of Capecitabine (Xeloda®) and Pegylated Interferon Alfa-2A(Pegasys®) for Recurrent or Progressive Brain Metastasis From Breast Carcinoma
Brief Title: Capecitabine and Pegylated Interferon Alfa-2a in Treating Patients With Recurrent or Progressive Brain Metastases Due to Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study slow to accrue.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0727; MDA-2004-0727; NCI-6810; CDR0000443592 (Other: NCI)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer; tumors metastatic to brain
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Breast Neoplasms, Male; Brain Neoplasms | interventions — peginterferon alfa-2a; Interferon alpha-2; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine + PEG-interferon alfa-2a (Experimental): Capecitabine 1000 mg/m2 orally twice daily during the first 14 days of each 3-week cycle (2 weeks on, 1 week rest), and PEG-interferon alfa-2a subcutaneously beginning at 180 mcg per week for 21 days.
  Interventions: Biological: PEG-interferon alfa-2a; Drug: Capecitabine

INTERVENTIONS:
Biological: PEG-interferon alfa-2a — Once a week subcutaneous injection for 21 days, beginning at 180 mcg per week. Repeated for additional 21 days to begin at the same time as repeat 21 day Capecitabine cycle.
  Other Names: PEGSYS; Interferon-alfa-2a; Interferon alpha 2a recombinant; Pegylated interferon alfa-2a
Drug: Capecitabine — 1000 mg/m^2 twice daily during first 14 days of each 3-week cycle (2 weeks on, 1 week rest).
  Other Names: Xeloda

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pegylated interferon alfa-2a may interfere with the growth of tumor cells. Giving capecitabine together with pegylated interferon alfa-2a may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine together with pegylated interferon alfa-2a works in treating patients with recurrent or progressive brain metastases due to breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of capecitabine and pegylated interferon alfa-2a, in terms of 6-month neurologic progression-free rate, in patients with recurrent or progressive brain metastases secondary to breast cancer.

Secondary

* Determine the toxicity spectrum of this regimen in these patients.
* Determine the time to neurologic progression and overall survival of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral capecitabine twice daily on days 1-14 and pegylated interferon alfa-2a subcutaneously on days 1, 8, and 15. Treatment repeats every 3 weeks for at least 6 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 38-98 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer that metastasized to the brain, meeting all of the following criteria:

  * Must have ≥ 1 inoperable brain metastases, meeting 1 of the following criteria:

    * Progressive or recurrent disease after prior whole-brain or stereotactic radiotherapy
    * Ineligible for OR unwilling to be treated with radiotherapy
  * At least 1 unidimensionally measurable brain metastasis by enhanced MRI within the past 21 days
  * No progression or development of central nervous system (CNS) metastasis during prior treatment with capecitabine, fluorouracil, interferon alfa, or interferon beta
* Systemic (i.e., outside the CNS system) cancer must be stable

  * No progressive disease (e.g., liver, lymphangitic, or lung metastases)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 mg/dL
* No history of idiopathic thrombocytopenic purpura
* No known uncontrolled coagulopathy
* No increased risk for anemia (e.g., thalassemia or spherocytosis)
* No medically problematic anemia

Hepatic

* aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) ≤ 2.5 times upper limit of normal (ULN) (5 times ULN for patients with concurrent liver metastases )
* Bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN for patients with concurrent liver metastases; 10 times ULN for patients with concurrent bone metastases)

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 30 mL/min

Cardiovascular

* No congestive heart failure
* No symptomatic coronary artery disease
* No medically uncontrolled arrhythmia
* No other clinically significant cardiac disease
* No myocardial infarction within the past 12 months

Gastrointestinal

* No history of inflammatory bowel disease
* Must have intact upper gastrointestinal tract
* Able to swallow tablets
* No malabsorption syndrome
* No history of gastrointestinal bleeding

Immunologic

* No prior unanticipated severe reaction to fluoropyrimidine therapy, interferon, pegylated interferon, or a pegylated moiety
* No known sensitivity to fluorouracil
* No serious uncontrolled infection
* No history of immunologically mediated disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No known dihydropyrimidine dehydrogenase deficiency
* No history of depression characterized by a suicide attempt
* No history of hospitalization for psychiatric disease
* No history of other severe psychiatric disease
* No prior disability as a result of psychiatric disease
* No history of clinically significant psychiatric disability that would preclude study compliance
* No other malignancy within the past 5 years except cured nonmelanoma skin cancer or treated carcinoma in situ of the cervix
* No uncontrolled thyroid dysfunction (e.g., thyroid-stimulating hormone not in normal range)
* No evidence of severe retinopathy (e.g., Cytomegalovirus (CMV) retinitis or macular degeneration)
* No clinically relevant ophthalmologic disorders due to diabetes or hypertension
* No other serious uncontrolled medical conditions that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 3 months since prior interferon alfa or interferon beta

Chemotherapy

* See Disease Characteristics
* At least 3 months since prior capecitabine or fluorouracil

Endocrine therapy

* Concurrent hormonal agents (e.g., tamoxifen, raloxifene, or anastrazole) for breast cancer allowed

Radiotherapy

* See Disease Characteristics

Surgery

* More than 4 weeks since prior major surgery and recovered

Other

* More than 4 weeks since prior participation in another investigational drug study
* At least 4 weeks since prior and no concurrent brivudine or sorivudine
* No concurrent cimetidine
* No other concurrent investigational or commercial agents or therapies for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Neurologic progression-free survival rate at 6 months | 6 months

SECONDARY OUTCOMES:
Time to neurologic progression | 6 months or until disease progression
Overall survival | Up to 2 years
Tumor response (complete response and partial response) | 6 months
  Response Evaluation Criteria in Solid Tumors (RECIST) criteria for Target (Brain Metastasis) Lesions where Complete Response (CR): Disappearance of all target lesions; and Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Toxicity | 6 months
  Toxicity defined as grade 3 or 4 hematologic, skin (hand and foot syndrome), or fatigue/myalgia/flu debilitation-syndrome (interferon-related) toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Groves, MD, JD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Cancer Research for the Ozarks, Springfield, Missouri
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas